CLINICAL TRIAL: NCT00160667
Title: An Exploratory, Double Blind, Randomized, Placebo-controlled, Parallel Group, Multicenter Study, for the Assessment of Efficacy, Safety and Tolerability of Ucb 34714 50 mg Oral Capsules in b.i.d. Administration at the Doses of 200 mg/Day and 400 mg/Day, in Subjects (at Least 18 Years Old) Suffering From Post Herpetic Neuralgia (PHN)
Brief Title: A Study Assessing Efficacy of Brivaracetam in Subjects With Persistent Pain After Shingles (Post-herpetic Neuralgia)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: UCB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01162; 2004-000975-32 (EudraCT Number)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Neuralgia, Postherpetic
Keywords: Post-herpetic Neuralgia (PHN); Brivaracetam
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo tablets administered twice a day.
  Interventions: Drug: Placebo
- Brivaracetam 200 mg/day (Experimental): Brivaracetam 200 mg/day (100 mg administered twice a day).
  Interventions: Drug: Brivaracetam
- Brivaracetam 400 mg/day (Experimental): Brivaracetam 400 mg/day (200 mg administered twice a day).
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Placebo — Daily oral dose of two equal intakes.
  Arms: Placebo
Drug: Brivaracetam — Daily oral dose of two equal intakes.
  Other Names: Briviact
  Arms: Brivaracetam 200 mg/day; Brivaracetam 400 mg/day

SUMMARY:
Study will assess efficacy, safety and tolerability of brivaracetam in post-herpetic neuralgia (PHN). Duration of 7 weeks divided into 3 periods with no up-titration, nor down-titration.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Male/female subject aged 18 years or older.
* Pain present for at least 6 months after healing of the acute herpes zoster skin rash.
* Pain intensity score assessed on an 11-point numerical pain rating scale with a score of at least 4 at the screening visit and with an average weekly score of at least 4 on an 11-point numerical pain rating scale during baseline period.

Exclusion Criteria:

* Subject getting any kind of psychological support to help cope with pain such as biofeedback or behavioral cognitive therapy.
* Subject who had undergone or who is scheduled for neurolytic or neurosurgical therapy for post-herpetic neuralgia (PHN) or who receives trans-electrical neural stimulation (TENS.
* Tricyclic antidepressants (TCAs) or non-steroidal anti-inflammatory drug (NSAIDs) or permitted opioid analgesics ('strong' opioids are forbidden) that started less than 30 days and/or are not stabilized prior to screening and/or are not expected to be kept stable during the study.
* Intake of more than two pain treatments at trial entry (screening visit) including Tricyclic antidepressants (TCAs), non-steroidal anti-inflammatory drugs (NSAIDs) or permitted opioid analgesics.
* Subject being treated with Carbamazepine for any indication.
* Known coexistent source of painful peripheral neuropathy or other systemic disease associated with a secondary painful neuropathy.
* Subject being treated in the four weeks prior to screening visit with 'strong' opioid analgesics.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2004-10-11 (Actual); Primary Completion 2006-01-05 (Actual); Study Completion 2006-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (50):
- Belgium (5):
  - Brussels
  - Eeklo
  - Genk
  - Liège
  - Lubbeek (Pellenberg)
- Bulgaria (3):
  - Pleven
  - Sofia
  - Varna
- Czechia (4):
  - Hradec Králové
  - Prague
  - Svitavy
  - Ústí nad Labem
- France (5):
  - Annecy
  - Clermont-Ferrand
  - Nice
  - Toulouse
  - Voiron
- Germany (5):
  - Bad Wörishofen
  - Bochum
  - Essen
  - Kassel
  - Rodgau
- Poland (11):
  - Gdansk
  - Grudziądz
  - Katowice
  - Kielce
  - Krakow
  - Lublin
  - Olsztyn
  - Poznan
  - Warsaw
  - Wroclaw
  - Zgierz
- Serbia (3):
  - Belgarde
  - Belgrade
  - Kragujevac
- Slovakia (4):
  - Bratislava
  - Dubnica nad Váhom
  - Košice
  - Nitra
- Spain (6):
  - Cadiz
  - Granada
  - Hospitalet de Llobregat (Barcelona)
  - Madrid
  - Sant Cugat Del Valles (Barcelona)
  - Valencia
- United Kingdom (4):
  - Bath
  - Glasgow
  - London
  - Winchester

REFERENCES:
- See also: Product Information — https://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in October 2004 and concluded in January 2006.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Period: Overall Study
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Started | 50 | 51 | 51
Completed | 45 | 48 | 45
Not Completed | 5 | 3 | 6
Not completed — Adverse Event | 3 | 1 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Patient decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to the Intention-to-treat (ITT) Set.
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day | Total Title
Number analyzed (Participants) | 50 | 51 | 51 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 22 | 23 | 62
  >=65 years | 33 | 29 | 28 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.06 (10.80) | 65.33 (10.95) | 65.58 (10.21) | 65.65 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 30 | 87
  Male | 21 | 23 | 21 | 65

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Average Pain Intensity Score From Baseline to the Last Week of the 4-week Treatment Period
Description: Pain intensity was scored on a 11-point numeric pain rating scale, ranging from 0 to 10 where 0= no pain and 10= worst possible pain.
  A negative value in percent change from Baseline indicates a decrease in average pain intensity score from Baseline.
Time Frame: Baseline, last week of the 4-week Treatment Period
Population: Only subjects with valid data for average pain intensity score at Baseline and the last week of the 4-week Treatment Period are included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 48 | 51 | 51
percentage of change | -26.16 (30.20) | -26.11 (33.73) | -27.36 (34.58)
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 200 mg/Day; Test type: Superiority or Other; p = 0.965, ANCOVA; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-12.82 to 13.41] — Estimated value is the difference of Least Square Means
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 400 mg/Day; Test type: Superiority or Other; p = 0.825, ANCOVA; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [-11.69 to 14.65] — Estimated value is the difference of Least Square Means

2. Secondary Outcome: Responder Rate in Average Pain Intensity Score at the Last Week of the Treatment Period Compared to the Baseline Period
Description: A responder is defined as a subject with a >= 30 % reduction in average pain intensity score at the Evaluation Week (last week of the Treatment Period) compared to the Baseline Period.
Time Frame: Baseline, last week of the 4-week Treatment Period
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 48 | 51 | 50
percentage of participants | 33.3 | 37.3 | 40.0

3. Secondary Outcome: Percent Change From the Baseline Period to Each Weekly Mean in the Pain Intensity Score
Description: as for outcome 1
Time Frame: Baseline, each Evaluation visit (up to Week 4)
Population: Intention-To-Treat set included 50 subjects treated with Placebo, 51 subjects treated with brivaracetam (BRV) 200 mg/day, 51 subjects treated with BRV 400 mg/day. Only subjects with valid data for pain intensity score at the respective visit (week) are included in the analysis. Number of participants analyzed is given separately per visit (week).
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 50 | 51 | 51
percentage of change
  Week 1: number analyzed (Participants) | 49 | 51 | 50
  Week 1 | -10.3 (13.8) | -5.2 (27.0) | -8.5 (20.2)
  Week 2: number analyzed (Participants) | 46 | 49 | 48
  Week 2 | -20.8 (26.4) | -10.5 (25.6) | -18.7 (22.0)
  Week 3: number analyzed (Participants) | 46 | 49 | 47
  Week 3 | -24.3 (29.3) | -20.2 (36.6) | -25.5 (29.2)
  Week 4: number analyzed (Participants) | 46 | 48 | 47
  Week 4 | -27.5 (29.6) | -25.8 (37.2) | -29.1 (33.7)

4. Secondary Outcome: Percent Change From the Baseline Period to the Last Week of the Treatment Period in the Sleep Interference Score
Description: Sleep interference was scored on a 11-point numerical sleep interference rating scale, ranging from 0 to 10 where 0 = 'pain does not interfere with sleep', 10 = 'pain completely interferes with sleep'.
  A negative value in percent change from Baseline indicates a decrease in average sleep interference score from Baseline.
Time Frame: Baseline, last assessment during the 4-week Treatment Period
Population: Only subjects with valid data for Sleep Interference Score are included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 42 | 48 | 46
percentage of change | -42.00 (37.41) | -23.33 (51.34) | -30.17 (59.27)

5. Secondary Outcome: Percent Change From the Baseline Period to Each Weekly Mean of the Treatment Period in the Sleep Interference Score
Description: as for outcome 4
Time Frame: Baseline, each Evaluation visit (up to Week 4)
Population: ITT set included 50 subjects treated with Placebo, 51 subjects treated with brivaracetam (BRV) 200 mg/day, 51 subjects treated with BRV 400 mg/day. Only subjects with valid data for Sleep Interference Score at the respective visit (week) are included in the analysis. Number of participants analyzed is given separately per visit (week).
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 50 | 51 | 51
percentage of change
  Week 1: number analyzed (Participants) | 43 | 48 | 46
  Week 1 | -13.06 (23.83) | -6.96 (28.63) | -18.01 (45.27)
  Week 2: number analyzed (Participants) | 40 | 46 | 44
  Week 2 | -33.28 (35.27) | -5.69 (46.43) | -27.38 (49.76)
  Week 3: number analyzed (Participants) | 40 | 46 | 43
  Week 3 | -34.75 (38.22) | -12.86 (55.79) | -35.46 (55.88)
  Week 4: number analyzed (Participants) | 40 | 45 | 43
  Week 4 | -42.92 (36.37) | -22.05 (54.92) | -37.60 (55.77)

6. Secondary Outcome: Absolute Change From the Randomization Visit to the Evaluation / Early Discontinuation Visit in the Total Pain Score of the Short-Form McGill Pain Questionnaire (SF-MPQ)
Description: The SF-MPQ has three components: the first one consists of 15 subscales (descriptors: 11 sensory, 4 affective) which are rated on an intensity scale with 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total subscales (descriptors). The SF-MPQ also includes a Present Pain Intensity (PPI) index and a visual analogue scale (VAS). Each of the 15 subscales is rated from 0=none to 3=severe pain. The Total Pain Score of the SF-MPQ is the sum of all 15 ratings and can hence vary from 0 (15*0=0: no pain) to 60 (15*4=60: severe pain). The mean change in total score is reported.
Time Frame: Randomization visit, Evaluation / Early Discontinuation visit (up to Week 4)
Population: Only subjects having values at randomization and at evaluation (V5) / early discontinuation are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 31 | 24 | 35
units on a scale | -3.44 (5.92) | -4.65 (6.80) | -4.62 (6.71)

7. Secondary Outcome: Absolute Change From the Randomization Visit to the Evaluation / Early Discontinuation Visit in the Sensory Score of the Short-Form McGill Pain Questionnaire (SF-MPQ)
Description: The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
  The sensory score ranges from 0 to 33. Change = observation mean at Evaluation / Early Discontinuation visit minus Randomization mean.
  A negative value in absolute change indicates an improvement.
Time Frame: Randomization visit, Evaluation / Early Discontinuation visit (up to Week 4)
Population: Only subjects having values at randomization and at Evaluation (V5) / Early Discontinuation are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 31 | 24 | 35
units on a scale | -2.42 (5.10) | -3.79 (5.50) | -4.17 (5.05)

8. Secondary Outcome: Absolute Change From the Randomization Visit to the Evaluation / Early Discontinuation Visit in the Affective Score of the Short-Form McGill Pain Questionnaire (SF-MPQ)
Description: The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
  The affective score ranges from 0 to 12. Change = observation mean at Evaluation / Early Discontinuation visit minus Randomization mean.
  A negative value in absolute change indicates an improvement.
Time Frame: Randomization visit, Evaluation / Early Discontinuation visit (up to Week 4)
Population: Only subjects having values at randomization and at evaluation (V5) / early discontinuation are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 31 | 23 | 36
units on a scale | -1.04 (2.16) | -0.70 (2.08) | -0.75 (3.07)

9. Secondary Outcome: Absolute Change From the Randomization Visit to the Evaluation / Early Discontinuation Visit in the Present Pain Intensity (PPI) Score of the SF-MPQ
Description: Present pain intensity (PPI) was rated by the subject. The score ranges from 0 (no pain) to 5 (excruciating). A negative value in absolute change indicates an improvement in PPI.
Time Frame: Randomization visit, Evaluation / Early Discontinuation visit (up to Week 4)
Population: Only subjects having values at randomization and at evaluation (V5) / early discontinuation are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 31 | 27 | 38
units on a scale | -0.7 (1.0) | -0.6 (1.3) | -0.9 (1.1)

10. Secondary Outcome: Absolute Change From the Randomization Visit to the Evaluation / Early Discontinuation Visit in the Visual Analog Scale (VAS) of the SF-MPQ
Description: Pain burden was rated by the subject using the visual analog scale (VAS) ranging from 0 (no pain) to 100 (worst possible pain). A negative value in absolute change indicates an improvement in pain burden.
Time Frame: Randomization visit, Evaluation / Early Discontinuation visit (up to Week 4)
Population: Only subjects having values at randomization and at evaluation (V5) / early discontinuation are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 33 | 27 | 38
units on a scale | -13.1 (27.2) | -15.5 (25.2) | -17.9 (31.8)

11. Secondary Outcome: Percentage of Subjects With Categorized Change in Pain Assessed by Patient's Global Evaluation Scale at the Evaluation / Early Discontinuation Visit
Description: Patient´s global assessment of change in pain was performed using a seven-point scale (7= Marked improvement, 6= Moderate improvement, 5= Slight improvement, 4= No change, 3= Slight worsening, 2= Moderate worsening, 1= Marked worsening).
Time Frame: Randomization visit, Evaluation / Early Discontinuation visit (up to Week 4)
Population: Only subjects with valid data at the Evaluation / Early Discontinuation visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 47 | 51 | 47
percentage of participants
  Marked improvement | 14.9 | 9.8 | 23.4
  Moderate improvement | 29.8 | 27.5 | 27.7
  Slight improvement | 12.8 | 25.5 | 10.6
  No change | 34.0 | 31.4 | 29.8
  Slight worsening | 6.4 | 5.9 | 6.4
  Moderate worsening | 2.1 | 0 | 2.1
  Marked worsening | 0 | 0 | 0

12. Secondary Outcome: Percentage of Subjects With Categorized Change in Post-herpetic Neuralgia Assessed by Investigator's Global Evaluation Scale at the Evaluation / Early Discontinuation Visit
Description: Investigator´s global assessment of change was performed using a seven-point scale (7= Marked improvement, 6= Moderate improvement, 5= Slight improvement, 4= No change, 3= Slight worsening, 2= Moderate worsening, 1= Marked worsening).
Time Frame: Randomization visit, Evaluation / Early Discontinuation visit (up to Week 4)
Population: Only subjects with valid data at the Evaluation / Early Discontinuation visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 49 | 51 | 51
percentage of participants
  Marked improvement | 10.2 | 9.8 | 17.6
  Moderate improvement | 28.6 | 23.5 | 23.5
  Slight improvement | 22.4 | 27.5 | 17.6
  No change | 34.7 | 39.2 | 27.5
  Slight worsening | 2.0 | 0 | 13.7
  Moderate worsening | 2.0 | 0 | 0
  Marked worsening | 0 | 0 | 0

13. Secondary Outcome: Percent Change From Randomization Visit to the Evaluation / Early Discontinuation in the Brush-evoked Allodynia Intensity Rated by the Patient
Description: Brush-evoked allodynia intensity was assessed by the subject on an 11-point numerical rating scale, ranging from 0= no pain to 10= unbearable Pain.
  A negative value in percent change indicates an improvement in brush-evoked allodynia intensity.
Time Frame: Randomization visit, Evaluation / Early Discontinuation visit (up to Week 4)
Population: Only subjects with valid data at the Evaluation / Early Discontinuation visit are included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 28 | 37 | 28
percentage of change | -27.4 (34.8) | -12.9 (39.3) | -18.2 (70.6)

14. Secondary Outcome: Percent Change From Randomization Visit to the Evaluation / Early Discontinuation in the Brush-evoked Allodynia Area Measured by the Investigator
Description: Allodynia is pain due to a normally non-painful stimulus. The brush-evoked allodynia areas were assessed by the Investigator (location and contour of the allodynic regions drawn on a standard dermatomal map). Areas (mm²) of the allodynic regions drawn by the Investigator were afterwards computed by means of appropriate tools and calibrated templates. The larger the area in square centimeters the more allodynia. A negative value in percent change in the brush-evoked allodynia area indicates improvement.
Time Frame: Randomization visit, Evaluation / Early Discontinuation visit (up to Week 4)
Population: Only subjects with valid data at the Evaluation / Early Discontinuation visit are included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
Number analyzed (Participants) | 5 | 9 | 10
percentage of change | -5.39 (17.18) | -25.18 (32.10) | 6.88 (92.50)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first intake of randomized study medication until Final Visit (Week 6)
Description: Adverse Events refer to the Safety Population consisting of all subjects who were dispensed medication.
Arm/Group | Placebo | Brivaracetam 200 mg/Day | Brivaracetam 400 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51 | 1/51
Other Adverse Events (participants affected / at risk) | 8/50 | 19/51 | 18/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | Brivaracetam 200 mg/Day (N=51) | Brivaracetam 400 mg/Day (N=51)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Vascular purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | Brivaracetam 200 mg/Day (N=51) | Brivaracetam 400 mg/Day (N=51)
Vertigo (Ear and labyrinth disorders) | 1 | 7 | 3
Nausea (Gastrointestinal disorders) | 1 | 1 | 4
Asthenia (General disorders) | 1 | 3 | 1
Fatigue (General disorders) | 2 | 3 | 6
Dizziness (Nervous system disorders) | 4 | 5 | 5
Headache (Nervous system disorders) | 1 | 4 | 2
Somnolence (Nervous system disorders) | 2 | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days